CLINICAL TRIAL: NCT02399163
Title: Clinical Evaluation of Oral Hygiene Products in an In Situ Caries Model
Brief Title: Evaluation of Oral Hygiene Products in an In Situ Caries Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 203160
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo dentifrice/Fluoride rinse (Experimental): Twice daily brushing with a non-fluoride (placebo) toothpaste followed by once daily rinsing (post night time brushing) with a fluoride mouthwash containing 220 ppm of fluoride as sodium fluoride
  Interventions: Drug: Fluoride free toothpaste; Drug: Fluoride mouthwash
- Placebo dentifrice/No rinse (Placebo Comparator): Twice daily brushing with a non-fluoride (placebo) toothpaste
  Interventions: Drug: Fluoride free toothpaste
- Fluoride dentifrice/No rinse (Active Comparator): Twice daily brushing with a fluoride toothpaste containing 1150 ppm of fluoride as sodium fluoride
  Interventions: Drug: Fluoride toothpaste
- Fluoride dentifrice/Fluoride rinse (Experimental): Twice daily brushing with a fluoride toothpaste containing 1150 ppm of fluoride as sodium fluoride, followed by once daily rinsing (post night time brushing) with a fluoride mouthwash containing 220 ppm of fluoride as sodium fluoride.
  Interventions: Drug: Fluoride toothpaste; Drug: Fluoride mouthwash

INTERVENTIONS:
Drug: Fluoride free toothpaste — Brushing with fluoride free toothpaste
  Arms: Placebo dentifrice/Fluoride rinse; Placebo dentifrice/No rinse
Drug: Fluoride toothpaste — Brushing with fluoride containing toothpaste
  Arms: Fluoride dentifrice/Fluoride rinse; Fluoride dentifrice/No rinse
Drug: Fluoride mouthwash — Fluoride mouth wash to be followed after brushing with fluoride free toothpaste in "Placebo dentifrice/Fluoride rinse" arm and in "Fluoride dentifrice/Fluoride rinse" arm
  Arms: Fluoride dentifrice/Fluoride rinse; Placebo dentifrice/Fluoride rinse

SUMMARY:
The study will evaluate and compare the potential anti-caries efficacy of a test regimen: placebo (fluoride free) toothpaste (twice daily use) plus fluoride mouthwash (once daily use), in comparison with brushing with a placebo toothpaste alone (twice daily use), to remineralize previously demineralized enamel specimens, as measured by Surface MicroHardness Recovery (%SMHR).

This will be a single center, randomized, laboratory analyst blinded, placebo, four treatment, cross-over study in healthy participants. Participants will be assessed at baseline and at the beginning and end of each treatment visit to monitor clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 85 years inclusive
2. Understands and is willing, able and likely to comply with all study procedures and restrictions
3. Good general and mental health with, in the opinion of the investigator or medically qualified designee:

   * No clinically significant and relevant abnormalities in medical history or upon oral examination.
   * Absence of any condition that could affect the participant's safety or well-being or their ability to understand and follow study procedures and requirements
4. Currently living in the Indianapolis, Indiana area and has not had a professional fluoride treatment within 14 days of the first treatment visit
5. Currently wearing a removable mandibular partial denture with sufficient room in one posterior buccal flange areas to accommodate two enamel specimens
6. Willing to have their denture modified to accommodate enamel test specimens and willing and capable of wearing their removable mandibular partial dentures 24 hours per day during the experimental periods
7. Have a salivary flow rate in the range of normal values (un-stimulated whole saliva flow rate ≥ 0.2 milliliter (mL)/minute; gum base stimulated whole saliva flow rate ≥ 0.8 mL/minute).

Exclusion Criteria:

1. Pregnant or breast feeding women
2. Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
3. Currently taking antibiotics or have taken antibiotics in the two weeks prior to the screening visit.
4. Taking or have taken a bisphosphonate drug for treatment of osteoporosis.
5. Participation in another GSKCH investigational dental product study within seven days of first study treatment.
6. Previous participation in this study.
7. Recent history (within the last year) of alcohol or other substance abuse.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center in United States of America.
Pre-assignment Details: A total of 80 participants were screened. Of the 80 participants, 62 were randomized and 53 completed the study.
Groups:
- Overall Study: In this cross-over study, participants were randomized to receive each of following treatments:
  1. Fluoride dentifrice/Fluoride rinse
  2. Placebo dentifrice/Fluoride rinse
  3. Fluoride dentifrice/No rinse
  4. Placebo dentifrice/No rinse
Period: Overall Study
Arm/Group | Overall Study
Started | 62
Completed | 53
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Protocol Deviation | 2
Not completed — Withdrawal by Participant | 5

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: All randomized participants were evaluated for baseline characteristics
Arm/Group | Overall Participants
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 30
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Surface Microhardness Recovery (%SMHR) of Placebo Dentifrice/Fluoride Rinse Compared to Placebo Dentifrice/No Rinse
Description: SMHR test was used to assess the changes in mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMHR was performed ex-vivo and determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents re-hardening of enamel surface. % SMH recovery was calculated from indentation length (micrometer [μm]) of sound enamel specimen at baseline(B), indentation length (μm) after in vitro demineralization(D1), indentation length (μm) after intra-oral exposure (R): [D1-R/D1-B]*100.
Time Frame: Baseline to 14 days
Population: Per-protocol (PP) population included all participants who were randomized into the study, received at least one dose of study product, had at least one post-baseline efficacy assessment and had no protocol violations deemed to affect efficacy during the study.
Measure: Mean (Standard Deviation); unit: % SMHR
Groups:
- Placebo Dentifrice/Fluoride Rinse: Twice daily brushing with a non-fluoride (placebo) toothpaste followed by once daily rinsing (post night time brushing) with a fluoride mouthwash containing 220 parts per million (ppm) of fluoride as sodium fluoride
Arm/Group | Placebo Dentifrice/Fluoride Rinse | Placebo Dentifrice/No Rinse
Number analyzed (Participants) | 53 | 52
% SMHR | 24.48 (16.088) | 8.09 (25.892)
Statistical Analysis 1: Comparison: Placebo Dentifrice/Fluoride Rinse vs Placebo Dentifrice/No Rinse; Test type: Superiority or Other; p < 0.0001, ANCOVA — From ANOVA: participant (random), treatment (fixed), period (fixed); Mean Difference (Net) = 16.76, 95% CI 2-sided [11.061 to 22.454] — Difference is Placebo dentifrice/Fluoride rinse minus Placebo dentifrice/No rinse such that a positive difference implies a larger response value for the Placebo dentifrice/Fluoride rinse

2. Secondary Outcome: Percentage Surface Microhardness Recovery (SMHR) of Placebo Dentifrice/Fluoride Rinse, Placebo Dentifrice/No Rinse, Fluoride Dentifrice/No Rinse and Fluoride Dentifrice/Fluoride Rinse
Description: SMHR test was used to assess the changes in mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMHR was performed ex-vivo and determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents rehardening of enamel surface. % SMH recovery was calculated from indentation length (micrometer [μm]) of sound enamel specimen at baseline(B), indentation length (μm) after in vitro demineralization(D1), indentation length (μm) after intra-oral exposure (R): [D1-R/D1-B]*100.
Time Frame: Baseline to 14 days
Population: PP population included all participants who were randomized into the study, received at least one dose of study product, had at least one post-baseline efficacy assessment and had no protocol violations deemed to affect efficacy during the study.
Measure: Mean (Standard Deviation); unit: % SMHR
Arm/Group | Placebo Dentifrice/Fluoride Rinse | Placebo Dentifrice/No Rinse | Fluoride Dentifrice/No Rinse | Fluoride Dentifrice/Fluoride Rinse
Number analyzed (Participants) | 53 | 52 | 54 | 52
% SMHR | 24.48 (16.088) | 8.09 (25.892) | 28.36 (21.037) | 30.01 (18.203)

3. Secondary Outcome: Enamel Fluoride Uptake
Description: The microdrill enamel biopsy technique was used to analyze the fluoride uptake by enamel. Each enamel specimen was mounted on the long axis of a drill attached to a microdrill and drilled to a depth of approximately 100 micrometer (μm) through the entire lesion (four cores per specimen). The enamel powder pooled from four drilling samples was then immediately analyzed for fluoride content using fluoride specific electrode and pH/ion meter. The amount of fluoride-uptake by enamel was calculated based on the amount of fluoride divided by the area of the enamel cores and expressed as microgram per square centimeter (μg/cm^2).
Time Frame: Baseline to 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram per square centimeter(μg/cm^2)
Arm/Group | Placebo Dentifrice/Fluoride Rinse | Placebo Dentifrice/No Rinse | Fluoride Dentifrice/No Rinse | Fluoride Dentifrice/Fluoride Rinse
Number analyzed (Participants) | 53 | 52 | 54 | 52
microgram per square centimeter(μg/cm^2) | 7.22 (3.016) | 1.60 (0.670) | 8.01 (3.925) | 9.97 (4.962)

4. Secondary Outcome: Change in Saliva Fluoride Concentration From Baseline (Pre-treatment) to Day 14
Description: Fluoride concentration in saliva was measured after collecting saliva samples at the following time points: - at Day 1 baseline prior to supervised treatment. - at day 1 post supervised treatment at site. - at Day 14 post treatment. The amount of fluoride in the samples was calculated based on the amount of fluoride divided by the volume of the sample and expressed as μg/mL of sample.
Time Frame: Baseline to Day14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram per mililitre(μg/mL )
Arm/Group | Placebo Dentifrice/Fluoride Rinse | Placebo Dentifrice/No Rinse | Fluoride Dentifrice/No Rinse | Fluoride Dentifrice/Fluoride Rinse
Number analyzed (Participants) | 53 | 51 | 54 | 52
microgram per mililitre(μg/mL ) | 0.06 (0.317) | -0.01 (0.030) | 0.00 (0.245) | 0.06 (0.203)

5. Secondary Outcome: Change in Saliva Fluoride Concentration From Baseline (Post-treatment) to Day 14
Description: Fluoride concentration in saliva was measured after collecting saliva samples at the following time points: - at Day 1 post supervised treatment at site. - at Day 14 post treatment. The amount of fluoride in the samples was calculated based on the amount of fluoride divided by the volume of the sample and expressed as μg/mL of sample.
Time Frame: Baseline up to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Placebo Dentifrice/Fluoride Rinse | Placebo Dentifrice/No Rinse | Fluoride Dentifrice/No Rinse | Fluoride Dentifrice/Fluoride Rinse
Number analyzed (Participants) | 53 | 51 | 54 | 52
μg/mL | 13.08 (9.743) | 0.05 (0.045) | 8.62 (6.892) | 13.81 (10.620)

ADVERSE EVENTS:
Arm/Group | Placebo Dentifrice/Fluoride Rinse | Placebo Dentifrice/No Rinse | Fluoride Dentifrice/No Rinse | Fluoride Dentifrice/Fluoride Rinse
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/56 | 0/59 | 1/57
Other Adverse Events (participants affected / at risk) | 15/60 | 13/56 | 18/59 | 17/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Dentifrice/Fluoride Rinse (N=60) | Placebo Dentifrice/No Rinse (N=56) | Fluoride Dentifrice/No Rinse (N=59) | Fluoride Dentifrice/Fluoride Rinse (N=57)
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Dentifrice/Fluoride Rinse (N=60) | Placebo Dentifrice/No Rinse (N=56) | Fluoride Dentifrice/No Rinse (N=59) | Fluoride Dentifrice/Fluoride Rinse (N=57)
Glossodynia (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Tongue Geographic (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip Dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral Discomfort (Gastrointestinal disorders) | 1 | 4 | 1 | 1
Paraesthesia Oral (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Tongue Ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival Erythema (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Gingival Hypertrophy (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival Oedema (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival Ulceration (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Lip Ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ORAL MUCOSAL ERYTHEMA (Gastrointestinal disorders) | 1 | 1 | 1 | 0
TRAUMATIC OCCLUSION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 1 | 1
ORAL HERPES (Infections and infestations) | 0 | 1 | 1 | 1
BRONCHITIS (Infections and infestations) | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 1 | 0
MOUTH INJURY (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
TONGUE INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
INJURY ASSOCIATED WITH DEVICE (General disorders) | 0 | 1 | 2 | 1
CHEST PAIN (General disorders) | 0 | 0 | 1 | 0
MEDICAL DEVICE PAIN (General disorders) | 1 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
SMEAR CERVIX ABNORMAL (Investigations) | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 2 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.